CLINICAL TRIAL: NCT02513420
Title: Perineal Muscle Training Versus Usual Prenatal Care in the Incidence of Avulsion of the Levator Ani Muscle at First Birth of Mexican Women: Randomized Control Trial
Brief Title: Levator Ani Muscle Avulsion at First Birth of Mexican Women: Randomized Control Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Daniel Velez Sanchez, Medical specialist, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: R-2014-3504-56
Record Dates: First submitted 2015-07-29; First posted 2015-07-31 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Trauma
Keywords: levator ani avulsion; perineal muscle training; pelvic floor ultrasound
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Perineal muscle training (Experimental): This group will recibe a training of a combination of perineal massage and pelvic floor muscle excersice that will start after 33 weeks of gestation. Every week until the childbith, They will be evaluated with a diary.
  Interventions: Behavioral: Perineal muscle training
- Usual prental care (No Intervention): Usually pregnant women have not a training focused in pelvic floor muscle, so this group won't receive any indication of pelvic floor training except if They complains of urinary incontinence.

INTERVENTIONS:
Behavioral: Perineal muscle training — It is a combination of perineal massage and Kegel exercises.
  Arms: Perineal muscle training

SUMMARY:
Levator Ani Muscle (LAM) avulsion occurs in 13-36% of women having their first birth. These damages by palpation and ultrasound of the pelvic floor can be detected. Avulsion of the LAM results in decreased muscle strength of the pelvic floor, enlarge the genital hiatus and promotes pelvic organ prolapse. The perineal muscle training is a proposal to combine the perineal massage with pelvic floor exercises in order to prepare the LAM in the last weeks before delivery, to withstand stretching which will be submitted during childbirth. No studies in the world that have explored the effect of the perineal muscle training on the avulsion of MEA.

Objective: To quantify the proportion of primiparous that result with avulsion of LAM after their first birth among those performing perineal muscle training from week 33 of gestation and those with usual prenatal care.

DETAILED DESCRIPTION:
This study will be performed in 228 primiparous. Previous informed consent they will be randomized in two groups: 1) perineal muscle training and 2) usual prenatal care. Pelvic floor will be evaluated before and after childbirth clinically and ultrasonographilly. The outcome variables will be: 1) avulsion LAM diagnosed by palpation and 2-3D pelvic floor ultrasound, 2) symptoms of pelvic floor dysfunction identified with standardized and validated Spanish PFDI-20 questionnaire, 3) changes dimension of the genital hiatus and perineal body, 4) accomplishment of perineal muscle training. Demographic variables (marital status, occupation, level of education, age, weeks of gestation, weight, height, BMI, religion, pathologies) and variables related to childbirth (weeks of gestation duration of the second period, use of analgesia, variety of position, episiotomy, forceps. dystocia, who attended the birth, weight and head circumference of the newborn, tearing report and who repairs the last one.

ELIGIBILITY:
Inclusion Criteria:

1. Future primiparous over 18 who have single fetus, without contraindications to take delivery. Primigesta omit the term since in the study patients who have had previous pregnancies that are not related to damage to the pelvic floor as will be accepted: abortions, ectopic or molar.
2. With or without symptoms of pelvic floor dysfunction (assessed with PFDI-20 questionnaire).
3. Have 33 weeks gestation to start participating, so the invitation must be made before this gestational age as mentioned above.
4. Physical and mental ability to understand and perform the maneuvers used in the study.

Exclusion Criteria:

1. Any contraindication to labor, this feature can appear at any time during pregnancy, including during labor.
2. Physical or mental inability to perform the maneuvers used in the study.
3. Avulsion of MEA detected before birth.
4. Agree not participate in the study.
5. Previous pregnancies older than 20 weeks gestation resolved abdominally.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-02-01 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Levator ani muscle avulsion | six weeks after childbith
  Lack of insertion of levator ani muscle to pubis identified by pelvic floor ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Vélez, M.Sc., Principal Investigator — Colegio Mexicano de Ginecología y Obstetricia
Locations (1):
- Instituto Mexicano del Seguro Social Centro Médico Nacional La Raza, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Krofta L, Otcenasek M, Kasikova E, Feyereisl J. Pubococcygeus-puborectalis trauma after forceps delivery: evaluation of the levator ani muscle with 3D/4D ultrasound. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1175-81. doi: 10.1007/s00192-009-0837-6. Epub 2009 Jul 29. PMID 19639235
- [Background] Albrich SB, Laterza RM, Skala C, Salvatore S, Koelbl H, Naumann G. Impact of mode of delivery on levator morphology: a prospective observational study with three-dimensional ultrasound early in the postpartum period. BJOG. 2012 Jan;119(1):51-60. doi: 10.1111/j.1471-0528.2011.03152.x. Epub 2011 Oct 10. PMID 21985531
- [Background] Schwertner-Tiepelmann N, Thakar R, Sultan AH, Tunn R. Obstetric levator ani muscle injuries: current status. Ultrasound Obstet Gynecol. 2012 Apr;39(4):372-83. doi: 10.1002/uog.11080. PMID 22190408
- [Background] DeLancey JO, Kearney R, Chou Q, Speights S, Binno S. The appearance of levator ani muscle abnormalities in magnetic resonance images after vaginal delivery. Obstet Gynecol. 2003 Jan;101(1):46-53. doi: 10.1016/s0029-7844(02)02465-1. PMID 12517644
- [Background] Kearney R, Miller JM, Ashton-Miller JA, DeLancey JO. Obstetric factors associated with levator ani muscle injury after vaginal birth. Obstet Gynecol. 2006 Jan;107(1):144-9. doi: 10.1097/01.AOG.0000194063.63206.1c. PMID 16394052
- [Background] Kearney R, Sawhney R, DeLancey JO. Levator ani muscle anatomy evaluated by origin-insertion pairs. Obstet Gynecol. 2004 Jul;104(1):168-73. doi: 10.1097/01.AOG.0000128906.61529.6b. PMID 15229017
- [Background] Lien KC, Mooney B, DeLancey JO, Ashton-Miller JA. Levator ani muscle stretch induced by simulated vaginal birth. Obstet Gynecol. 2004 Jan;103(1):31-40. doi: 10.1097/01.AOG.0000109207.22354.65. PMID 14704241
- [Background] Hoyte L, Damaser MS, Warfield SK, Chukkapalli G, Majumdar A, Choi DJ, Trivedi A, Krysl P. Quantity and distribution of levator ani stretch during simulated vaginal childbirth. Am J Obstet Gynecol. 2008 Aug;199(2):198.e1-5. doi: 10.1016/j.ajog.2008.04.027. Epub 2008 Jun 2. PMID 18513684
- [Background] Svabik K, Shek KL, Dietz HP. How much does the levator hiatus have to stretch during childbirth? BJOG. 2009 Nov;116(12):1657-62. doi: 10.1111/j.1471-0528.2009.02321.x. Epub 2009 Sep 1. PMID 19735376
- [Derived] Woodley SJ, Lawrenson P, Boyle R, Cody JD, Morkved S, Kernohan A, Hay-Smith EJC. Pelvic floor muscle training for preventing and treating urinary and faecal incontinence in antenatal and postnatal women. Cochrane Database Syst Rev. 2020 May 6;5(5):CD007471. doi: 10.1002/14651858.CD007471.pub4. PMID 32378735